CLINICAL TRIAL: NCT00839813
Title: Efficacy of Yoga for Treatment-Resistant PTSD
Brief Title: Efficacy of Yoga for Treatment-Resistant Posttraumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Justice Resource Institute (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Bessel van der Kolk, MD, The Trauma Center at JRI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT003905-01A2 (NIH); R21AT003905-01A2 (NIH); 1R21AT003905-01A2 (NIH)
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Yoga; Posttraumatic Stress Disorder; PTSD; women's health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga (Experimental): 10 week trauma-sensitive yoga classes
  Interventions: Behavioral: Yoga
- Women's Health Education (No Intervention): 10 weeks of women's health education classes as an attentional control group

INTERVENTIONS:
Behavioral: Yoga — 10 weeks of a trauma-sensitive yoga class
  Arms: Yoga

SUMMARY:
The central question in this research proposal is: can a popular technique that specifically targets active mastery and improved affect regulation, yoga, which is utilized by approximately 4% of the US population each year (1), improve the constellation of PTSD symptoms, multiple somatic complaints, social and occupational impairment and high health care utilization that has been documented in hundreds of thousands of women in the US?

The Primary Aims of this study include the following:

1. To test the short-term and long-term effectiveness of 10 weeks of yoga for treating treatment-resistant PTSD and compare it with attention controls receiving Women's Health Education (WHE).
2. To assess the short-term and long-term effects of yoga on a) co-morbid conditions, b) quality of life, c) body awareness, d) health care utilization and e) heart rate variability (HRV), in comparison to an attention control group.

DETAILED DESCRIPTION:
Research has demonstrated a close association between trauma exposure and 1) PTSD, anxiety & depression, 2) loss of affect regulation, 3) poor quality of life, and 4) high health care utilization (2, 3). This study will explore how a popular body-mind technique, yoga, compares with a attentional control group condition, Women's Health Education (WHE), in the treatment of [heretofore treatment- unresponsive adults with] PTSD, and measure whether yoga can affect "the attitudes and beliefs" that "can reduce psychological stress and contribute to positive health outcomes." [The study of yoga for chronic PTSD is in line with the empirical research that supports the notion that autonomic dysregulation plays a significant role in the persistence of PTSD (4), and with the hypothesis that an increased capacity for self-regulation is associated with a decrease in the severity of this symptom constellation].

Primary aims.

1. To test the short-term and long-term effectiveness of 10 weeks of yoga for treating treatment-resistant PTSD and compare it with attention controls receiving Women's Health Education (WHE).
2. To assess the short-term and long-term effects of yoga on a) co-morbid conditions, b) quality of life, c) body awareness, d) health care utilization and e) heart rate variability (HRV), in comparison to an attention control group.

Primary Hypotheses:

1. Participants in the yoga condition will demonstrate a clinically significant reduction in PTSD symptoms at post-treatment, defined as a mean reduction of total CAPS score of at least 30% compared to baseline.
2. Yoga will be more effective than attention control at improving PTSD symptoms as evidenced by a significantly greater drop in total CAPS score from pre-treatment to post-treatment for the yoga group.

   Secondary Hypotheses:
3. Yoga will be more effective at improving comorbid conditions and quality of life and reducing health care utilization than attention control.
4. Yoga will be more effective than attention control at improving HRV and body awareness.]

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 58 years old, any race
* Chronic, treatment-unresponsive PTSD
* An index trauma that occurred 12 or more years before initial interview
* At least 3 years of prior treatment focused on dealing with the consequences of the index trauma
* Comorbid diagnoses of depression or panic disorder, which are common in subjects with PTSD, will be permitted

Exclusion Criteria:

* Medical: Serious illness (including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease) that is not stabilized based on the judgment of the PI.
* Psychological: GAF < 40.
* Bipolar disorders, obsessive-compulsive disorder [OCD], schizophrenia, and any psychotic disorder will be excluded if they occurred any time prior to the primary traumatic episode
* Current psychotic disorder, or established organic impairment (e.g., TBI)
* Severe dissociation, as measured by a DES score >25.
* Women with active suicidal risk, active self-mutilation or aggressive behavior toward others within the past year, as judged by the PI
* Substance dependence or abuse in the past 6 months, as defined by DSM IV criteria and judged by the PI.
* Any other condition that might interfere with the person's capacity to give informed consent, or to adhere to the study protocol.
* Legal and Financial: Current legal proceedings resulting from the traumatic events. People whose continued receipt of financial benefits is contingent upon maintaining PTSD symptoms or who are waiting for a decision concerning the receipt of financial benefits based upon PTSD symptoms
* Prior Yoga Experience: Subjects who have attended more than five prior yoga sessions.

Ages: 18 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS 1) | Initial Assessment
Clinician Administered PTSD Scale (CAPS 1) | One week Pre-Treatment Evaluation
Clinician Administered PTSD Scale (CAPS 1) | One week Post-treatment
Clinician Administered PTSD Scale (CAPS 1) | 2 month-follow-up Evaluation

SECONDARY OUTCOMES:
Heart Rate Variability | Initial Assessment, week 1 of treatment, week 2 of treatment, week 5 of treatment, week 9 of treatment, week 10 of treatment, one week post-treatment, 2 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bessel van der Kolk, M.D., Principal Investigator — The Trauma Center at JRI
Locations (1):
- The Trauma Center at JRI, Brookline, Massachusetts, United States

REFERENCES:
- [Derived] Nguyen-Feng VN, Hodgdon H, Emerson D, Silverberg R, Clark CJ. Moderators of treatment efficacy in a randomized controlled trial of trauma-sensitive yoga as an adjunctive treatment for posttraumatic stress disorder. Psychol Trauma. 2020 Nov;12(8):836-846. doi: 10.1037/tra0000963. Epub 2020 Aug 27. PMID 32853015
- [Derived] van der Kolk BA, Stone L, West J, Rhodes A, Emerson D, Suvak M, Spinazzola J. Yoga as an adjunctive treatment for posttraumatic stress disorder: a randomized controlled trial. J Clin Psychiatry. 2014 Jun;75(6):e559-65. doi: 10.4088/JCP.13m08561. PMID 25004196